CLINICAL TRIAL: NCT03450798
Title: SOFT Block Versus Spinal Anesthesia in Patients Undergoing Surgery for Fixation of Open Tibial Fractures Using Ilizarov External Fixator
Brief Title: SOFT Block Versus Spinal Anesthesia in Patientsusing Ilizarov External Fixator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hoda Shokri, HShokri, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWA00001785
Record Dates: First submitted 2018-02-20; First posted 2018-03-01 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOFT block group (Active Comparator): needle will be introduced medial to the femoral vein and 3 cm below the skin where 15 mL of bupivacaine 0.25% injected. the obturator nerve, the probe shifted medially, superior to the needle, and directed cranially to the pectineus muscle . Needle withdrawn to the subcutaneous tissue and redirected using out-of-plane toward the deep surface of pectineus, 10 mL of bupivacaine 0.25%will be injected. The sciatic nerve, we use the curvilinear probe, inferior to the needle, and tilted the probe to get the clearest image of the sciatic nerve.The needle will be inserted then withdrawn subcutaneously and directed by an in-plane toward the sciatic nerve deep to the inferior border of the quadratus femoris muscle.20 mL of bupivacaine 0.25% will be injected
  Interventions: Device: SOFT block group
- spinal anesthesia group (Sham Comparator): patients will receive spinal anesthesia with hyperbaric bupivacaine 0.5% (7.5-10mg). This will be administered via a 25-G spinal needle at L4-L5 or L3-L4 with the patient in the sitting position under complete aseptic conditions.
  Interventions: Device: spinal anesthesia group

INTERVENTIONS:
Device: SOFT block group — needle will be introduced medial to the femoral vein and 3 cm below the skin where 15 mL of bupivacaine 0.25% injected. the obturator nerve, the probe shifted medially, superior to the needle, and directed cranially to the pectineus muscle . Needle withdrawn to the subcutaneous tissue and redirected using out-of-plane toward the deep surface of pectineus, 10 mL of bupivacaine 0.25%will be injected. The sciatic nerve, we use the curvilinear probe, inferior to the needle, and tilted the probe to get the clearest image of the sciatic nerve.The needle will be inserted then withdrawn subcutaneously and directed by an in-plane toward the sciatic nerve deep to the inferior border of the quadratus femoris muscle.20 mL of bupivacaine 0.25% will be injected
  Arms: SOFT block group
Device: spinal anesthesia group — patients will receive spinal anesthesia with hyperbaric bupivacaine 0.5% (7.5-10mg). This will be administered via a 25-G spinal needle at L4-L5 or L3-L4 with the patient in the sitting position under complete aseptic conditions.
  Arms: spinal anesthesia group

SUMMARY:
Peripheral nerve block is an ideal choice for lower limb surgery because of the peripheral site of the surgical procedure and the ability to block pain pathways at multiple levels. On the contrary to other anesthetic techniques, as spinal or general anesthesia, properly performed peripheral nerve blocks bypass adverse events as hemodynamic instability and respiratory complications, properly treat post-operative pain leading to early hospital discharge. Additional advantages of peripheral nerve blocks are that they can be used in patients receiving anti-coagulants or lumbosacral disease in addition to avoidance of airway instrumentation.

Recently, there has been a significant interest in regional anesthesia and peripheral nerve blockade. This is facilitated by a significant advance of the research in this field and availability of better equipment facilitating regional anesthesia.The aim of this study was to assess the efficacy and safety of SOFT block (sciatic-obturator-femoral nerve block technique) in comparison with spinal anesthesia in patients undergoing surgery for fixation of open tibial fractures using Ilizarov external fixator.

DETAILED DESCRIPTION:
After the approval of medical ethical committee of Ain Shams University, this prospective parallel group double blinded study will be conducted over 60 patients between the age of 35-57 years old, ASA physical status I and II, scheduled for fixation of open tibial fractures using iIlizarov external fixator. at Ain Shams University hospitals in 2018-2019, After written informed consent is obtained.

Refusal to participate, inability to communicate with the investigators or hospital staff, obesity (body mass index>40 kg/m2), patients undergoing bilateral surgery, patients with coagulopathies ,renal insufficiency (creatinine>1.5 mg/dL), American Society of Anesthesia (ASA) III-IV, patients with any contraindication to regional anesthesia , patients with unstable vital data and patients with head or chest trauma will be excluded.

Preanesthetic check will be done at night of surgery. After an intravenous (IV) cannula will be secured , and midazolam 0.05 mg/kg i.v. will be given to all patients before transfer to the operating room where standard monitoring devices as ECG,Non invasive blood pressure and pulse oximetry will be placed. Then, patients will be randomly allocated by sealed envelope technique to receive either spinal anesthesia or SOFT block. In spinal anesthesia group, patients will receive spinal anesthesia with hyperbaric bupivacaine 0.5% (7.5-10mg). This will be administered via a 25-G spinal needle at L4-L5 or L3-L4 with the patient in the sitting position under complete aseptic conditions.

In SOFT group, patients will receive SOFT block where patients will be positioned in supine position,under aseptic conditions, a linear US probe will be placed on the inguinal crease to show the femoral nerve and vessels. Using an in-plane technique, a 12-cm stimulating block needle will be introduced medial to the femoral vein and advanced 1-3 cm below and parallel to the skin. Then, It will be redirected toward the fibres of the femoral nerve, where 15 mL of bupivacaine 0.25% will be injected. To block the obturator nerve, the probe will be shifted medially, superior to the needle, and directed cranially to identify the pectineus muscle . The needle will be then withdrawn to the subcutaneous tissue and redirected using an out-of-plane technique toward the deep surface of the pectineus, where 10 mL of bupivacaine 0.25%will be injected.[4 ] To locate the sciatic nerve, we will use the curvilinear probe, directed it inferior to the needle, and tilted the probe to get the clearest image of the sciatic nerve.The needle will be inserted then withdrawn subcutaneously and directed by an in-plane technique toward the sciatic nerve deep to the inferior border of the quadratus femoris muscle. Then 20 mL of bupivacaine 0.25% will be injected after needle elicited muscle twitches using 1 mA current.

Sensory level will be evaluated by loss of pinprick sensation (20-gauge hypodermic needle).

Haemodynamic variables will be recorded every 5 min after block performance until the end of surgery. Hypotension will be defined as a decrease in systolic arterial blood pressure by 30% or more from baseline values, and it will be initially treated with 200 ml IV infusion of Ringer's lactate solution; if this proved to be ineffective, an IV bolus of phenylephrine (40-50 mcg) will be given. Bradycardia is defined as heart rate decrease below 45 bpm, and it was treated with 0.5 mg IV atropine.

Sensory block(loss of pinprick sensation at T12 in the Spinal group, or in the femoral, obturator and sciatic nerves distribution in the SOFT group). The quality of the block will be judged according to the need for supplementary IV analgesics and sedation: adequate nerve block = neither sedation nor analgesics required to complete surgery; inadequate nerve block = need for rescue dose of analgesic (100 mg IV bolus of ketamine) or sedation (3mg IV midazolam) will be required to complete surgery; failed nerve block so general anesthesia will be required to complete surgery.

After completion of surgery, patients will be transferred to the post-anesthesia care unit (PACU). Intravenous pethidine (50 mg) will be given as rescue analgesic as needed. Primary endpoint is the time from the end of local anaesthetic injection to complete resolution of sensory block. The secondary endpoints include patient satisfaction, (on a numerical rating scale), the adverse events as back pain, postural -puncture headache , vomiting, adverse events of systemic toxicity from local anesthetic as seizures and cardiovascular collapse, persistent parasthesia observed within 48 hours after the block and failure rate of the block will be recorded.

In case of failure of the block or incidence of seizures resulting from local anesthetic toxicity , we will convert to general anesthesia.

In case of cardiovascular collapse, support the patient with intravenous fluids and vasopressors as required so in these cases patients will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 57 years old
* ASA I,II
* BMI<30
* fixation of open tibial fractures using Ilizarov external fixator -

Exclusion Criteria:

* Refusal to participate,
* Inability to communicate with the investigators or hospital staff,
* body mass index>40 kg/m2
* patients undergoing bilateral surgery,
* History of coagulopathies
* creatinine>1.5 mg/dL
* American Society of Anesthesia (ASA) III-IV
* Any contraindication to regional anesthesia
* Unstable vital data
* Head or chest trauma will be excluded.

Ages: 35 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
T- test of the recovery time(duration of analgesia)mean±SD | 3-12 hours
  It is the time from the end of local anaesthetic injection to complete resolution of sensory block

SECONDARY OUTCOMES:
Review of medical records for postoperative complications | 48 hours after the procedure
  persistent parasthesia
Failure of the block | 50 minutes
  general anesthesia will be required to complete surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Shokri, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol
Time Frame: 5 to 6 months
Access Criteria: The collected data are coded, tabulated, and statistically analyzed using statistical package for social sciences software, version 17.0 (SPSS Inc., Chicago, Illinois, USA). Descriptive statistics are carried out for numerical parametric data and presented as mean±SD, whereas categorical data are presented as number and percentage. Variables such as demographic data and comorbidities are compared using the χ2-test. A P value less than 0.05 was considered significant.

REFERENCES:
- [Derived] Shokri H, Kasem AA. Sciatic obturator femoral technique versus spinal anaesthesia in patients undergoing surgery for fixation of open tibial fractures using Ilizarov external fixator. A randomised trial. BMC Anesthesiol. 2020 Jan 4;20(1):4. doi: 10.1186/s12871-019-0920-6. PMID 31901231